CLINICAL TRIAL: NCT03250585
Title: Secretory Phospholipases A2 in Exhaled Breath Condensate From Sickle Cell Patients With Acute Chest Syndrome: A Feasibility Study
Brief Title: sPLA2 in EBC During Acute Chest Syndrome
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: HM20010698
Record Dates: First submitted 2017-08-10; First posted 2017-08-15 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Sickle Cell Disease; Acute Chest Syndrome
Keywords: acute chest syndrome; secretory phospholipases A2; exhaled breath condensate; sickle cell disease
MeSH Terms: conditions — Anemia, Sickle Cell; Acute Chest Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sickle Cell Patients with Acute Chest Syndrome: Sickle cell patients with active acute chest syndrome (ACS) from which samples of EBC and plasma will be collected during acute illness within 48 hours of admission with or diagnosis of ACS (Time point 1) in 3 sessions each 1 hour apart (Time point 1a, 1b, and 1c), and 2 weeks after discharge when have returned to steady-state (Time point 2). Time point 2 samples will serve as control (baseline) samples.
  Interventions: Diagnostic Test: Exhaled Breath Condensate (EBC); Diagnostic Test: Plasma Sample

INTERVENTIONS:
Diagnostic Test: Exhaled Breath Condensate (EBC) — Serial EBC samples will be collected within 48 hours of acute chest syndrome (ACS) diagnosis and at 2 week follow up
Diagnostic Test: Plasma Sample — Serial plasma samples will be collected within 48 hours of acute chest syndrome (ACS) diagnosis and at 2 week follow up

SUMMARY:
Secretory phosholipases A2 (sPLA2) are significantly elevated in the plasma of sickle cell disease patients with acute chest syndrome (ACS), and similar enzymes have been measured in exhaled breath condensate (EBC), which is collected easily and non-invasively. The investigators hypothesize that sPLA2 will be measurable in EBC samples from sickle cell patients with acute chest syndrome.

DETAILED DESCRIPTION:
The purpose of this research study is to test the ease and effectiveness of collecting exhaled breath condensate (liquid) to measure levels of a biomarker, secretory phospholipases A2 (sPLA2) in people with sickle cell disease during an attack of acute chest syndrome. sPLA2 levels have been reported to be much higher in persons with acute chest syndrome and might be useful to diagnose and to evaluate the effects of therapy.

Serial monitoring of plasma sPLA2 levels might lead to earlier or more accurate detection of acute chest syndrome and monitoring of its progression or improvement in patients with sickle cell disease. However, there is a significant inherent risk of frequent blood collection further dropping the blood (hemoglobin) levels of an already anemic patient. If sPLA2 can be measured in exhaled breath condensate, this non-invasive and well-tolerated sample collection might allow for serial monitoring of the enzyme without depleting the patient's already diminished blood supply.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of sickle cell anemia (the most severe types of sickle cell disease) as demonstrated by one of the following genotypes: HbSS, HbSβ0
2. Age ≥ 7 and < 40 years
3. Diagnosis of ACS as defined below
4. EBC collection able to be initiated within 48 hours of diagnosis of ACS

Definition of acute chest syndrome to be used: New radiographic pulmonary infiltrate of at least one complete lung segment in addition to 2 or more of the following symptoms: fever, chest pain, dyspnea, tachypnea, hypoxia. Given the small number of subjects in this feasibility study, we are using the more conservative definition in order to ensure samples are from patients with true ACS. This will increase the likelihood that sPLA2 levels will be high enough for measurement.

Exclusion Criteria:

1. Blood product transfusion in the previous 3 months (due to potential alterations in biomarkers, including sPLA2)
2. Chronic inflammatory conditions other than sickle cell (due to elevation from baseline of sPLA2 in inflammatory conditions)
3. Physical inability to correctly breathe into the mouthpiece for the required amount of time without compromising respiratory status
4. Intubated patients (though EBC can be measured in intubated patients, we will not include this subpopulation for the purpose of this study)
5. Pregnancy (due to the hematologic and respiratory changes that physiologically occur during gestation)

Ages: 7 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Sickle cell patients with acute chest syndrome
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2018-06-14 (Actual); Study Completion 2018-06-14 (Actual)

PRIMARY OUTCOMES:
sPLA2 Measurement in EBC during ACS | Time point 1 (within either 48 hours of admission or time of diagnosis of ACS, if not present on admission)
  sPLA2 level in EBC at Time point 1 (during acute ACS episode) as measured by ELISA
sPLA2 Levels in EBC during ACS versus Steady-State | Time point 1 to Time point 2 (at 2 week follow-up)
  Comparison of sPLA2 levels in EBC from Time point 1 (during acute illness) and Time Point 2 (return to baseline status at 2 week follow up).

SECONDARY OUTCOMES:
sPLA2 levels in EBC versus Plasma | Time point 1 (within either 48 hours of admission or time of diagnosis of ACS, if not present on admission)]
  Difference in sPLA2 levels from EBC compared with Plasma during Time point 1 (during acute illness)

CONTACTS AND LOCATIONS:
Overall Officials: Davis D Michael, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States